CLINICAL TRIAL: NCT01191242
Title: Methadone Monitoring for Insights Into Adverse Events
Acronym: MEMORIES
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 154-08
Record Dates: First submitted 2010-08-17; First posted 2010-08-30 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2012-04

CONDITIONS: Pain; Opiate Addiction
Keywords: methadone; genetic
MeSH Terms: conditions — Pain; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Methadone has been an effective and inexpensive therapy in the management of chronic pain and opioid dependence. However it has been associated with sudden, unexpected deaths. Two mechanisms have been suggested, increased drug concentration in the blood, and a change in the heart rhythm. This study will look at blood samples for drug levels and genetic components and EKG's (a noninvasive test which reveals heart rhythm). There will be no intervention.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years of age or older; eligible for methadone treatment as judged by Discovery House criteria
* must sign informed consent for methadone treatment prior to being approached for this study
* must sign a written informed consent for this study
* is willing and has a means to return for all scheduled follow-up visits

Exclusion Criteria:

* pregnancy, participation in any other clinical trial involving investigational or marketed products with 30 days prior to entry into this study; current use of an inducer/inhibitor of known enzymes involved with methadone metabolism
* use of methadone in the 30 days prior to study enrollment; concomitant use of QT prolonging drugs
* considered by the treatment physician to be ineligible for methadone treatment; hepatic function panel indicates chronic liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects initiating methadone treatment for opioid addiction who meet elibitility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Carlquist, PhD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Discovery House, Taylorsville, Utah

REFERENCES:
- [Derived] Carlquist JF, Moody DE, Knight S, Johnson EG, Fang WB, Huntinghouse JA, Rollo JS, Webster LR, Anderson JL. A Possible Mechanistic Link Between the CYP2C19 Genotype, the Methadone Metabolite Ethylidene-1,5-Dimethyl-3,3-Diphenylpyrrolidene (EDDP), and Methadone-Induced Corrected QT Interval Prolongation in a Pilot Study. Mol Diagn Ther. 2015 Apr;19(2):131-8. doi: 10.1007/s40291-015-0137-4. PMID 25903311

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone Maintenance Observation Group: A consecutive sample of individuals initiating methadone maintenance treatment for opioid addiction.
Period: Overall Study
Arm/Group | Methadone Maintenance Observation Group
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 23
  Hispanic | 6
  African American | 1
  Native American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Total Methadone Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 107.3 (50.6)
  Day 7 | 315.4 (129.6)
  Day 21 | 362.2 (213.1)

2. Primary Outcome: Total Methadone Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 53.0 (27.3)
  Day 7 | 162.6 (68.5)
  Day 21 | 211.1 (119.5)

3. Primary Outcome: (S)- Methadone Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 65.6 (29.9)
  Day 7 | 178.8 (76.9)
  Day 21 | 215.1 (103.1)

4. Primary Outcome: (S)- Methadone Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 32.2 (14.4)
  Day 7 | 84.2 (39.5)
  Day 21 | 106.1 (60.1)

5. Primary Outcome: (R)-Methadone Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 41.8 (21.1)
  Day 7 | 136.6 (55.3)
  Day 21 | 178.6 (90.8)

6. Primary Outcome: (R)-Methadone Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 23.0 (11.8)
  Day 7 | 78.4 (31.8)
  Day 21 | 105.0 (61.4)

7. Primary Outcome: Total 2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidene (EDDP) Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 11.0 (8.6)
  Day 7 | 39.8 (33.4)
  Day 21 | 45.3 (27.0)

8. Primary Outcome: Total EDDP Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 4.8 (4.5)
  Day 7 | 17.7 (10.0)
  Day 21 | 26.6 (16.7)

9. Primary Outcome: (S)-EDDP Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 5.8 (3.8)
  Day 7 | 20.6 (15.5)
  Day 21 | 30.3 (19.0)

10. Primary Outcome: (S)-EDDP Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 3.8 (2.3)
  Day 7 | 9.1 (6.7)
  Day 21 | 13.7 (9.4)

11. Primary Outcome: (R)-EDDP Peak Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 3.4 (3.1)
  Day 7 | 13.5 (10.3)
  Day 21 | 18.2 (9.0)

12. Primary Outcome: (R)-EDDP Trough Plasma Concentration
Time Frame: Day 1, Day 7, Day 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Methadone Maintenance Observation Group
Number analyzed (Participants) | 31
ng/mL
  Day 1 | 1.2 (1.7)
  Day 7 | 6.6 (3.7)
  Day 21 | 10.5 (6.9)

ADVERSE EVENTS:
Description: All-cause mortality, serious, and other (not including serious) adverse events were not monitored/assessed.
Arm/Group | Methadone Maintenance Observation Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The principal limitations are small sample size and the limited number of genetic variants tested. Also, study endpoints were not examined beyond 21 days of treatment; thus the durability of study findings over longer time periods is not known.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes